CLINICAL TRIAL: NCT01843478
Title: A Test of an Intervention to Improve Pap Testing Among Women With HIV
Brief Title: The Self-Collection Study: a Study of Self-collected HPV Testing and Results Counseling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NA_00071156; F31NR013633-01 (NIH)
Record Dates: First submitted 2013-04-26; First posted 2013-04-30 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: HIV Infection
Keywords: women; human immunodeficiency virus; cervical cancer screening; Pap testing; human papillomavirus
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HPV Self-Collection (Experimental): The intervention is a self-collected HPV test, followed by results counseling by phone when the result is available (usually 2-3 weeks). Women are encouraged to have Pap testing.
  Interventions: Other: Self-Collected HPV Test
- Usual Care (Placebo Comparator): In the usual care arm, women do not receive the HPV test. They are encouraged to have Pap testing. In addition, there is a phone call as an attention control, where women are reminded to make a Pap test appointment about 2-3 weeks after the baseline visit.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Self-Collected HPV Test — The HPV self-collected test is followed by results counseling by phone when the result is available (usually 2-3 weeks). Women are encouraged to have Pap testing.
  Other Names: HPV test (Qiagen hc2)
  Arms: HPV Self-Collection
Other: Usual Care
  Arms: Usual Care

SUMMARY:
Cervical cancer is the second most common type of cancer among women worldwide. Women with human immunodeficiency virus (HIV) bear a disproportionate burden of cervical cancer and its precursor, cervical intraepithelial neoplasia (CIN), that result from persistent high-risk Human Papillomavirus (HPV) infection. HIV clinical practice guidelines recommend two Pap tests in the year following diagnosis, and if both are normal, yearly thereafter. Nationally, only 25% of women meet this recommendation. The mean annual Pap testing rate for federally funded HIV centers is only 55.7%. In 2009, quality improvement statistics from the Johns Hopkins Hospital Moore Clinic, a large urban HIV center, revealed an annual Pap testing rate of 59%. This occurred despite interventions to address adherence issues were implemented, including nurse case management, co-location of HIV and gynecology services, flexible scheduling, and continuity of care. Women keep their appointments for HIV primary care more often than for gynecology care in the Moore Clinic, so an intervention that takes place during a primary care visit could improve cervical cancer screening rates.

The availability of HPV testing provides a unique opportunity to increase perceived susceptibility to and severity of cervical cancer among women with HIV, and to encourage follow-up Pap testing. HPV testing involves analyzing a sample of cervicovaginal cells for the presence of high-risk HPV strains. Detection of high-risk strains of the virus indicates a high risk for high grade CIN and cancer, while a negative HPV test predicts a less than 2% risk of developing CIN. HPV testing can be easily conducted by women themselves through self-collection in a primary care visit. Studies of women without HIV who do not have regular Pap testing have demonstrated that self-collected HPV testing and results counseling increases the overall screening rate, and women who test positive for HPV have a high rate of follow-up Pap testing. Self-collected HPV testing and results counseling could be utilized in the HIV primary care setting to promote Pap testing among women with HIV.

DETAILED DESCRIPTION:
This study is a randomized trial to test whether receiving self-collected HPV testing and results counseling in HIV primary care will increase completion of Pap testing in a group of women attending the Johns Hopkins Hospital Moore Clinic for HIV Care. The study is informed by the Health Belief Model (HBM), which posits that screening behavior will increase if persons at risk for disease have a cue to action that increases their perception of susceptibility to and severity of the disease. In this study, the HPV test and results counseling are cues to action that also correctly identify those women at high risk for disease. To achieve these aims, 111 women who are late for Pap testing will be recruited for participation while they are at an HIV care appointment. They will be randomized to HPV self-collection and results counseling, or to receive usual care. Six months after enrollment, medical records will be reviewed for completion of Pap testing in the intervening months.

ELIGIBILITY:
Inclusion Criteria:

- HIV infection 18 months or more since Pap test Speak & read English Eligible for cervical cancer screening Plans to have Pap testing at Johns Hopkins Hospital

Exclusion Criteria:

- History of hysterectomy Currently pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Pap test | 6 months
  The outcome measure is the completion of Pap testing within 6 months of the baseline study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Hayley Mark, PhD, MPH, RN, Principal Investigator — Johns Hopkins University
Locations (1):
- Moore Clinic for HIV Care, Johns Hopkins Hospital, Baltimore, Maryland, United States